CLINICAL TRIAL: NCT04755205
Title: A Natural History Study of Children and Adults With Olfactory Neuroblastoma
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 210009; 21-C-0009
Record Dates: First submitted 2021-02-13; First posted 2021-02-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01-22

CONDITIONS: Olfactory Neuroblastoma; Esthesioneuroblastoma
Keywords: esthesioneuroblastoma; nasal cavity tumor; pediatric onb; adult onb; Natural History
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects with confirmed olfactory neuroblastoma.

SUMMARY:
Background:

Olfactory neuroblastoma (ONB) is a rare cancer. It grows from tissue in the upper part of the nose cavity, related to the sense of smell and can affect a person s sense of smell. Researchers want to better understand the health problems of people with ONB. This may help them design better treatment and supportive care studies.

Objective:

To better understand ONB-the course of the disease, tumor characteristics, response to treatments, and management of the treatment.

Eligibility:

People ages 3 years and older who have ONB. They must enroll in NIH studies #19-C-0016 and #18-DC-0051.

Design:

Participants will be screened with a medical history and medical record review.

Participants do not have to visit NIH.

Participants will give a blood sample. They will complete surveys to assess their emotional and physical wellbeing and needs. Leftover tissue from biopsies and surgeries will be collected.

Participants will take smell tests. They will smell items and answer questions about them.

Participants may take taste tests. They will get plastic taste strips that they will move around their mouth to determine the taste.

Participants may have a physical exam. Their performance status may be assessed.

Participants may give blood, saliva, urine, and nasal secretion samples.

Participants may have computed tomography and/or magnetic resonance imaging scans.

Participants may have one or more tumor biopsies.

Participants will talk to the research team about the results of their medical record/tests evaluation. The team will recommend how to best manage and treat their disease.

Participants may give samples and complete surveys every 12 months. Their medical records will be reviewed every year. They will be monitored for the rest of their life.

DETAILED DESCRIPTION:
Background:

Olfactory neuroblastoma (ONB), also known as esthesioneuroblastoma, is a malignant tumor of the nasal cavity believed to arise from the olfactory epithelium. ONB is rare, with a reported incidence of 0.4 per million (approximately 300 cases per year in the United States).

ONB most frequently arises in adults aged 20-60 years. Pediatric ONB is particularly rare, with only small case series or multi-institutional studies reported. However, a Surveillance Epidemiology and End Results (SEER) study of 47 pediatric patients with intranasal malignancy reported ONB as the most frequent pediatric intranasal malignancy (28%).

Due to the location of ONB in the sinonasal tract and anterior skull base, the presenting symptoms are often non-specific, including nasal obstruction and epistaxis, thus patients often present at advanced stages. Furthermore, ONB has a propensity for local invasion and relatively high rates of distant spread most commonly to the neck, lungs, and bones.

Clinical management in adults is generally surgical with adjuvant radiation.

The natural history of pediatric and adult ONB is incompletely understood, and treatment options for recurrent or metastatic ONB are limited. The planned natural history study as part of the NCI POB Rare Tumor Patient Engagement Network (RTPEN) will allow for comprehensive evaluation and recommendations to these patients while longitudinally collecting clinical, epidemiologic, and biological data.

Objective:

To characterize the natural history of ONB including clinical presentation, family history, patterns of disease progression, response to current treatment methods, disease recurrence, and overall survival

Eligibility:

Participants of age >= 3 years old with histologically documented ONB.

Design:

This protocol is intended to characterize the natural history of olfactory neuroblastoma.

Participants will undergo a comprehensive study entry evaluation including acquisition of imaging of tumor sites.

Medical histories will be documented, and participants followed throughout the course of their disease, with particular attention to patterns of disease recurrence and progression, response to therapies, duration of responses, and patient reported outcomes. Specimens will be obtained longitudinally, when feasible, and tumor growth rates will also be assessed throughout the course of the disease, when feasible.

Blood and tumor samples may be obtained at study entry and while on study.

ELIGIBILITY:
* INCLUSION CRITERIA:.
* Subjects with histologically documented olfactory neuroblastoma.
* Age >= 3 years old.
* Ability of subject to understand and the willingness to sign a written consent document

EXCLUSION CRITERIA:

Pregnant women are excluded from this study because of more than minimal risk activities (imaging studies with contrast, biopsies) pertaining to enrollment.

Ages: 3 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with olfactory neuroblastoma.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize the natural history of ONB | duration of study
  To characterize the natural history of ONB including clinical presentation, family history, patterns of disease progression, response to current treatment methods, disease recurrence, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0009.html